CLINICAL TRIAL: NCT05452811
Title: Open Retropubic Versus Laparoscopic Colposuspension (Burch Operation) Techniques for Female Stress or Mixed Urinary Incontinence; A Ten-year Experience in a Tertiary Center
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ozan Karadeniz, Principal investigator, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: KanuniSSSEAH
Record Dates: First submitted 2022-07-04; First posted 2022-07-11 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Stress Urinary Incontinence
Keywords: Burch colposuspension; laparoscopy; outcome; retropubic; stress urinary incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Open Burch Colposuspension: The retropubic space was entered through a laparotomy Pfannenstiel incision, and two permanent sutures were placed on each side lateral to the urethra, one set at the level of the mid urethra and the other set at the level of the bladder neck.
  Interventions: Procedure: Burch colposuspension
- Laparoscopic Burch Colposuspension: After a pneumo peritoneum was established entrance to the retropubic space began with a transverse incision of the anterior peritoneum using sharp dissection and electrocautery. The space was developed using blunt and sharp dissection to identify clearly the retropubic anatomy, including the pubic symphysis, bladder neck, and Cooper's ligaments. The bladder neck was identified and the paraurethral tissue was exposed. A no. 0 permanent suture then was introduced through the 10-mm port and was grasped with a laparoscopic needle driver. With the surgeon's hand in the vagina to elevate the paraurethral tissue, two figure-of-eight sutures incorporating full-thickness vagina excluding epithelium were placed on each side, one set lateral to the mid urethra and the other set lateral to the bladder neck. Each of these sutures then was passed through the ipsilateral Cooper's ligament and was secured with a series of extracorporeal knots using an endoscopic knot pusher.
  Interventions: Procedure: Burch colposuspension

INTERVENTIONS:
Procedure: Burch colposuspension — Anti-incontinence surgery for stress urinary incontinence

SUMMARY:
To evaluate postoperative course, efficacy, and complication rates of Open Burch Colposuspension and Laparoscopic Burch Colposuspension techniques in stress or mixed urinary incontinence at a single training and research hospital over the last 10 years in Istanbul, Turkey.

DETAILED DESCRIPTION:
A retrospective cohort study was conducted in all Burch Colposuspension cases performed between January 2001 and May 2022 at Kanuni Sultan Süleyman Training and Research Center. All patients' data were reviewed from the electronic medical records and analyzed who underwent Burch colposuspension surgery either with an open or laparoscopic approach. The primary outcome was surgical success, whereas secondary outcomes were perioperative and postoperative data including surgical type (open or laparoscopic), operating time, duration of hospital stay, estimated blood loss, complications during surgery, and additional interventional procedure types.

ELIGIBILITY:
Inclusion Criteria:

* patients having SUI or mixed urinary incontinence whom conservative therapy (Kegel's pelvic floor exercises, bladder training, electrical stimulation, or medication) failed
* SUI had been proven by urodynamic assessments.
* patients who had urethral hypermobility supported by a Q-type test with a cotton swab angle greater than 300
* patients having a residual urinary volume of less than 100 mL were included.

Exclusion Criteria:

* history of anti-incontinence surgery
* pelvic inflammatory diseases
* urinary retention
* SUI with intrinsic sphincter deficiency
* neurogenic bladder
* suspected malignancy
* urge incontinence
* chronic cystitis
* urinary tract infection
* prescription of anticoagulant or antipsychotic treatment
* coagulation disorders
* physically and medically unsuitable for colposuspension surgery
* pregnancy and loss to follow-up.

Min Age: 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A retrospective cohort study was performed on 150 patients with a diagnosis of SUI or mixed urinary incontinence who underwent anti-incontinence surgery between January 2011 to May 2022 in the department of Obstetrics and Gynecology of Kanuni Sultan Suleyman Training and Research Center in Istanbul.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Surgical success | 12 months after intervention
  Provided by the patient's feeling of the "Absence of a bulge in the vagina"

SECONDARY OUTCOMES:
estimated blood loss | intraoperative
  Blood loss during surgery ( taking blood count-WBC)
complications | up to 6 weeks
  Complications occurring in between during surgery and 6.th week of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No